CLINICAL TRIAL: NCT06958315
Title: An Observational Prospective Study to Assess the Effectiveness of Inclisiran(Leqvio®)in Patients With Atherosclerotic Vascular Disease and/or Heterozygous Familial Hypercholesterolemia Treated in Spanish Clinical Practice:the INSPIRE Study
Brief Title: Inclisiran (Leqvio®) in Patients With Atherosclerotic Vascular Disease and/or Heterozygous Familial Hypercholesterolemia Treated in Spain: the INSPIRE Study
Acronym: INSPIRE
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839A1ES03
Record Dates: First submitted 2025-04-25; First posted 2025-05-06 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Atherosclerotic Vascular Disease; Heterozygous Familial Hypercholesterolemia
Keywords: inclisiran; Leqvio®; atherosclerotic vascular disease; heterozygous familial hypercholesterolemia; Spanish clinical practice; Spain; INSPIRE; LDL-C goal attaiment
MeSH Terms: conditions — Atherosclerosis | interventions — ALN-PCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No samples will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inclisiran: Adults (≥18 years) with a confirmed clinical indication for inclisiran.
  Interventions: Other: Inclisiran

INTERVENTIONS:
Other: Inclisiran — This is an observational study, there is no treatment allocation.
  Other Names: KJX839 Leqvio

SUMMARY:
This study aims to address several key questions regarding the use of inclisiran in real-world clinical practice in Spain.

DETAILED DESCRIPTION:
The objective of the study is to determine the proportion of Atherosclerotic cardiovascular disease (ASCVD) and/or Heterozygous Familial Hypercholesterolemia (HeFH) patients reaching low-density lipoprotein-cholesterol (LDL-C) goals according to their cardiovascular risk at 12 months after the initiation of inclisiran treatment.

The study also aims to evaluate changes in LDL-C levels, safety profile, adherence and persistence to inclisiran treatment, use of concomitant lipid-lowering therapy (LLT), and patient satisfaction with inclisiran among other variables collected in clinical practice.

This is a non-interventional, prospective, multicentric, and nationwide study that will be conducted in routine clinical practice in Spain. This study will consist of three visits, coinciding with those conducted as part of the patients' routine follow-up, without interfering with the clinical practice of the participating centers. A blood test to assess LDL-C levels will be conducted at 3, 6, 9 and 12 months after inclisiran initiation, according to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years.
2. Written signed informed consent form (ICF).
3. Patients with a confirmed clinical indication for inclisiran who have received the first dose of inclisiran, following clinical judgement, at least 2 months prior to the inclusion in the study.
4. Available assessment of LDL-C levels (mg/dL) within 6 months before inclisiran initiation. The measurement of LDL-C levels must be done after one month of stable LLT and without any modification from the testing up to inclisiran initiation.
5. Statin-intolerant patients are eligible if they had documented side effects on ≥2 statins, including one at the lowest dose.

Exclusion Criteria:

1. Participating in a clinical trial of a treatment that could modify LDL-C levels during the observational period of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with a confirmed clinical indication for inclisiran.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
LDL-C levels - 12 months | 12 months following the initiation of inclisiran treatment.
  Proportion of participants reaching guideline-established low densitiy lipoprotein-Cholesterol (LDL-C) targets according to their Cardiovascular (CV) risk
  * LDL-C <55 mg/dL for ASCVD participants.
  * LDL-C <70 mg/dL for HeHF patients.

SECONDARY OUTCOMES:
LDL-C levels - 6 months | 6 months following the initiation of inclisiran treatment
  Proportion of participants reaching guideline-established LDL-C targets according to their CV risk
  * LDL-C <55 mg/dL for ASCVD participants.
  * LDL-C <70 mg/dL for HeHF patients.
non-HLDL-C levels | 6 and 12 months following the initiation of inclisiran treatment
  Proportion of participants with hypertriglyceridemia (triglycerides >400 mg/dL) reaching guideline-established non-HDL-C targets according to their CV risk
  * Non-HDL-C <85 mg/dL for ASCVD patients.
  * Non-HDL-C <100 mg/dL for HeHF patients.
Changes from baseline in LDL-C | Baseline, 3, 6, 9 and 12 months following the initiation of inclisiran treatment
  Change from baseline to mean LDL-C in PCSK9i naïve patients and patients pre-treated with PCSK9i, separately.
Frequency of AEs | From inclisiran initiation up to 12 months post-initiation
  Incidence of AEs including, number of cardiovascular events, revascularizations, emergency visits, and hospitalizations qualifying and reported as AEs.
Adherence rate to the concomitant LLT treatment | From 1st visit up to 12 months after inclisiran initiation
  Number of participants with a Morisky Medication Adjerence Slace (MMAS) of over 80%To describe the utilization and adherence to concomitant LLT during inclisiran treatment.
Proportion of participants adhering to the prescribed inclisiran dosing schedule | From 1st visit up to 12 months after inclisiran initiation
  To evaluate treatment adherence to inclisiran during the study period.
Inclisiran reasons for non-persistence | From 1st visit up to 12 months after inclisiran initiation
  Number of participants by reasons for non- persistence
Lp(a) | When available, from baseline up to 12 months after inclisiran initiation
  Proportion of participants with Lp(a) ≥50 mg/dL (≥125 nmol/L), ≥70 mg/dL (≥175 nmol/L), ≥90 mg/dL (≥225 nmol/L).
Changes in Lp(a) | From inclisiran initiation up to 12 months post-initiation
  To describe changes in Lp(a) at any time after inclisiran treatment, only in patients tested by clinical judgment.
Patient satisfaction with inclisiran, score on TSQM-II | 3 and at 12 months after treatment initiation.
  Treatment Satisfaction Questionnaire for Medication II evaluates satisfaction with treatment effectiveness, side effects, convenience, and global satisfaction. The TSQM-II consists of 11 items, each with 7 response options. Scores for each domain are calculated by averaging responses, transformed to a 0-100 scale, where higher scores indicate greater satisfaction
Specialty of the health care profesional prescribing inclisiran | From 1st visit up to 12 months after inclisiran initiation
  To describe prescribing specialty.
HCP who administers inclisiran | From 1st visit up to 12 months after inclisiran initiation
  To describe, HCP that administer inclisiran
Site of treatment administration for each dose | From 1st visit up to 12 months after inclisiran initiation
  To describe site of treatment administration (primary, secondary or tertiary hospital, primary care center)

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - Novartis Investigative Site, Cadiz, Andalusia
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Huelva, Andalusia
  - Novartis Investigative Site, Jaén, Andalusia
  - Novartis Investigative Site, Marbella, Andalusia
  - Novartis Investigative Site, Puerto Real, Cadiz
  - Novartis Investigative Site, Logroño, La Rioja
  - Novartis Investigative Site, Burgos
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Fuerteventura
  - Novartis Investigative Site, Las Palmas GC
  - Novartis Investigative Site, León
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com/